CLINICAL TRIAL: NCT06859918
Title: ASPE Subproject - Training to Understand and Navigate Emotions and Interactions (TUNE In)
Brief Title: Randomized Clinical Trial of TUNE In 3.0: A Social/Emotional Program for Adults With Autism Spectrum Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TUNE In 3.0
Record Dates: First submitted 2025-02-27; First posted 2025-03-05 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Autism Spectrum Disorder; Autism; Autistic Disorder; Asperger Syndrome
Keywords: Social Skills; Emotion Regulation; Autistic Adults
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder; Asperger Syndrome; Social Skills; Emotional Regulation | interventions — Drug Interactions

STUDY DESIGN:
Intervention Model Description: This study involves two groups of participants, who both receive the intervention at different times. The "Immediate Start Group" will get the intervention at the beginning of the trial, while the "Delay Start Group" will receive the intervention 1-6 months after the Immediate Start Group. Participants will be randomly assigned to groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Delay Start Group (Other): The Delay Start Group receives the intervention 1-6 months after the Immediate Start Group.
  Interventions: Behavioral: TUNE In: Training to Understand and Navigate Emotions and Interactions
- Immediate Start Group (Experimental): The Immediate Start Group receives the intervention as soon as the trial starts.
  Interventions: Behavioral: TUNE In: Training to Understand and Navigate Emotions and Interactions

INTERVENTIONS:
Behavioral: TUNE In: Training to Understand and Navigate Emotions and Interactions — A cognitive behavioral treatment strategy to improve social functioning in adults with autism spectrum disorder. TUNE In includes components to address the many behavioral domains involved in social functioning, including social motivation, social anxiety, social cognition, and social skills.

SUMMARY:
The purpose of this study is to test a novel, cognitive behavioral treatment strategy to improve social functioning in adults with autism spectrum disorder.

The treatment, named TUNE In (Training to Understand and Navigate Emotions and Interactions), includes components to address the many behavioral domains involved in social functioning, including social motivation, social anxiety, social cognition, social skills, and generalization of the skills to community settings.

The Investigators will test the efficacy of TUNE In to improve social functioning in adults with autism spectrum disorder (ASD), using a randomized controlled trial using the SRS-2 as the primary outcome measure.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Meet ASD diagnostic criteria supported by an outside diagnostic evaluation and/or by the clinical and developmental information gathered from a phone screen
* Be willing to complete screening surveys (outcome measures)
* Social Responsiveness Score, Second Edition, self-report SRS survey score of greater than or equal to 60

Exclusion Criteria:

* Severe self-injurious or aggressive behaviors; or with suicidal or homicidal ideation or behaviors (e.g. suicide attempt) within the last 6 months
* Major mood episode (major depressive episode, manic episode), psychotic symptoms, or a psychiatric hospitalization within the last 6 months
* A history of intellectual disability or low Shipley-2 score

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03-24 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Social Responsiveness Scale (SRS) - Self Report | From enrollment to 6 months follow up
  A 65 item self-report measure that identifies the presence and severity of social impairment within the autism spectrum.

SECONDARY OUTCOMES:
Social Responsiveness Scale (SRS) - Informant Report | From enrollment to 6 months follow up
  A 65 item measure that identifies the presence and severity of social impairment within the autism spectrum. This is completed by a friend/family member of the participant based on their perceptions of the participants' behavior.
CAT-Q - Camouflaging Autistic Traits Questionnaire | From enrollment to 6 months follow up
  A 25 item measure that assesses the extent to which individuals with autism mask or camouflage their autistic traits in social situations.
Five Facet Mindfulness Questionnaire | From enrollment to 6 months follow up
  A 39-item measure that assesses five aspects of mindfulness: observing, describing, acting with awareness, non-judging, and non-reactivity.
Generalized Anxiety Disorder-7 | From enrollment to 6 months follow up
  A 7-item measure that assesses the severity of generalized anxiety disorder symptoms.
Glasgow Sensory Questionnaire | From enrollment to 6 months follow up
  A 42-item measure that assesses sensory sensitivities and differences across multiple sensory modalities.
Insomnia Severity Inde | From enrollment to 6 months follow up
  A 7-item measure that assesses the severity of insomnia symptoms and their impact on daily functioning.
Inventory of Socially Supportive Behaviors | From enrollment to 6 months follow up
  A 40-item measure that assesses the frequency and types of social support individuals receive.
Social Network Index | From enrollment to 6 months follow up
  A 12-item measure that assesses the size, diversity, and level of engagement in an individual's social network.
Scales of Psychological Wellbeing | From enrollment to 6 months follow up
  A 42 item measure that assesses six dimensions of psychological well-being: autonomy, environmental mastery, personal growth, positive relations with others, purpose in life, and self-acceptance.
Attunement Quiz | From enrollment to 6 months follow up
  A 25 item measure that assess attunement: one's ability to perceive, interpret, and respond to one's internal and external environment, in particular the social environment.
Liebowitz Social Anxiety Scale - Self-Report | From enrollment to 6 months follow up
  A 24-item measure that assesses the severity of social anxiety symptoms related to fear and avoidance in social and performance situations.

CONTACTS AND LOCATIONS:
Overall Officials: Edward Brodkin, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Brodkin Lab: Perelman School of Medicine, Department of Psychiatry, University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be available through NIH NDAR registry
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Deidentified data will be uploaded to NDAR upon completion of the trial